CLINICAL TRIAL: NCT01253811
Title: A Multi-Centre, Multinational, Open-Label, Single-Arm and Multiple Dosing Trial on Safety and Efficacy of Monthly Replacement Therapy With Recombinant Factor XIII (rFXIII) in Paediatric Subjects With Congenital Factor XIII A-subunit Deficiency. Safety Extension Trial to F13CD-3760
Brief Title: Safety and Efficacy of Monthly Replacement Therapy With Recombinant Factor XIII (rFXIII) in Paediatric Subjects With Congenital Factor XIII A-subunit Deficiency
Acronym: mentor™5
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F13CD-3835; U1111-1117-1063 (Other: WHO); 2010-020192-23 (EudraCT Number)
Record Dates: First submitted 2010-12-01; First posted 2010-12-03 (Estimated); Results first posted 2016-06-24 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-05

CONDITIONS: Congenital Bleeding Disorder; Congenital FXIII Deficiency
MeSH Terms: interventions — recombinant factor XIII-A2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- rFXIII 35 IU/kg (Experimental)
  Interventions: Drug: catridecacog

INTERVENTIONS:
Drug: catridecacog — Intravenous injection of a single dose of recombinant factor XIII, 35 IU/kg body weight every 4th week
  Other Names: recombinant factor XIII

SUMMARY:
This trial will be conducted in Asia, Europe and the United States of America (USA).

The aim of this clinical trial is to investigate long-term safety of rFXIII when administered for prevention of bleeding episodes in children aged between 1 and 6 years with congenital FXIII A-subunit deficiency. This trial is an extension to trial F13CD-3760 (mentor™4, NCT01230021). If applicable the trial will be extended up to maximum 3 years dependent on when recombinant factor XIII will be commercially available in subject's respective country for use in children of 1-6 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Completed participation in trial F13CD-3760 (NCT01230021)

Exclusion Criteria:

* Known or suspected hypersensitivity to trial product or related products
* Known history of development of inhibitors against FXIII (factor XIII)
* Hereditary or acquired coagulation disorder other than FXIII congenital deficiency
* Platelet count (thrombocytes) less than 50X10e9 / L
* Previous history of autoimmune disorder involving autoantibodies e.g., systemic lupus erythematosus
* Previous history of arterial or venous thromboembolic events e.g., cerebrovascular accident or deep vein thrombosis
* Any disease or condition which, judged by the trial physician, could imply a potential hazard to the subject, interfere with the trial participation or trial outcome including renal and/or liver dysfunction

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2011-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (4):
- United States (2):
  - Novo Nordisk Clinical Trial Call Center, Boston, Massachusetts
  - Novo Nordisk Clinical Trial Call Center, Columbus, Ohio
- Petah Tikva, Israel
- Leicester, United Kingdom

REFERENCES:
- [Derived] Kerlin BA, Inbal A, Will A, Williams M, Garly ML, Jacobsen L, Kearney SL. Recombinant factor XIII prophylaxis is safe and effective in young children with congenital factor XIII-A deficiency: international phase 3b trial results. J Thromb Haemost. 2017 Aug;15(8):1601-1606. doi: 10.1111/jth.13748. Epub 2017 Jul 10. PMID 28581691
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 5 sites in 3 countries as follows: Israel (IS): 1 site; United Kingdom (UK): 2 sites; and United States (US): 2 sites.
Pre-assignment Details: Subjects who completed the F13CD-3760 (NCT01230021) trial were eligible to get enrolled in this trial.
Groups:
- rFXIII 35 IU/kg: Subjects received 35 IU/kg recombinant factor XIII (rFXIII) slow intravenous (i.v.) administered every 4 weeks (28 ± 2 days) as preventive treatment of bleeding episodes. Each dose was reconstituted, diluted with saline and injection was given at a rate not exceeding 1-2 mL min-1. This dose was identical to the dose administered in the trial F13CD-3760. The correct dosing was calculated based on subject's body weight. Subjects received rFXIII either at the clinic during the first year or as home treatment after one year, and only if allowed, according to local regulations.
Period: Overall Study
Arm/Group | rFXIII 35 IU/kg
Started | 6
Exposed | 6
Completed | 5
Not Completed | 1
Not completed — Withdrawal criteria | 1

BASELINE CHARACTERISTICS:
Population: The safety analysis set (SAS) included all patients exposed to trial drug (rFXIII).
Arm/Group | rFXIII 35 IU/kg
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.0 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment Emergent (Serious and Non-serious) Adverse Events
Description: An adverse event was described as any untoward medical occurrence in a subject or clinical investigation subject administered a pharmaceutical product, and which does not necessarily have a causal relationship with this treatment. Treatment emergent adverse events (serious and non-serious), defined as adverse events occurring from first trial product administration to the end of the subject's participation in the trial.
Time Frame: Week 0 to end of trial visit (week 173) for a minimum period of 52 weeks.
Population: The safety analysis set included all subjects who received at least one dose of the trial product.
Measure: Number; unit: number of events
Arm/Group | rFXIII 35 IU/kg
Number analyzed (Participants) | 6
number of events
  All adverse events | 100
  Serious adverse events | 2
  Non-serious adverse events | 98

2. Secondary Outcome: Percentage of Subjects With Development of Anti-rFXIII Antibodies, Including Inhibitors.
Description: All subjects who received rFXIII were monitored for the frequency of development of anti-rFXIII antibodies. Samples passed through 2 tiers of ELISA testing: an initial screen with a specific cut-off point (including ~5% false positives) and a second confirmatory assay for samples yielding a result above the screening cut-off point. If samples were confirmed as antibody positive in the confirmation assay, an inhibitor assay was also carried out to detect functional inhibitors.
Time Frame: Week 0 to end of trial visit (week 173).
Population: The SAS included all subjects who received at least one dose of the trial product. There were no antibodies against rFXIII detected in any patient during the trial.
Measure: Number; unit: percentage of subjects
Arm/Group | rFXIII 35 IU/kg
Number analyzed (Participants) | 6
percentage of subjects | 0

3. Secondary Outcome: Clinical Laboratory Assessments: Biochemistry: Creatinine
Description: Clinical laboratory assessments for creatinine at week 24 to end of trial visit.
Time Frame: Every 6th month, from week 24 to end of trial visit (week 173).
Population: The safety analysis set included all subjects who received at least one dose of the trial product.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | rFXIII 35 IU/kg
Number analyzed (Participants) | 6
mmol/L
  Week 24 (pre-dose), N=5 | 30.20 (8.23)
  Week 48 (pre-dose), N=5 | 28.00 (6.16)
  Week 72 (pre-dose), N=6 | 28.67 (5.13)
  Week 96 (pre-dose), N=5 | 37.00 (4.74)
  Week 120 (pre-dose), N=4 | 31.50 (5.92)
  Week 144 (pre-dose), N=3 | 31.00 (6.00)
  Week 168 (pre-dose), N=1 | 55.00 (0.00)
  End of trial (week 173) pre-dose, N= 6 | 35.17 (9.79)

4. Secondary Outcome: Clinical Laboratory Assessments: Biochemistry: Urea
Description: Clinical laboratory assessments for urea at week 24 to end ot trial visit.
Time Frame: Every 6th month, week 24 to end of trial visit (week 173).
Population: The safety analysis set included all subjects who received at least one dose of the trial product.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | rFXIII 35 IU/kg
Number analyzed (Participants) | 6
mmol/L
  Week 24 (pre-dose), N=5 | 5.50 (1.63)
  Week 48 (pre-dose), N=5 | 4.00 (1.22)
  Week 72 (pre-dose), N=6 | 3.99 (0.69)
  Week 96 (pre-dose), N=5 | 4.50 (1.14)
  Week 120 (pre-dose), N=4 | 3.48 (0.73)
  Week 144 (pre-dose), N=3 | 4.52 (1.35)
  Week 168 (pre-dose), N=1 | 5.00 (0.00)
  End of trial (week 173) pre-dose, N= 6 | 4.28 (0.84)

5. Secondary Outcome: Clinical Laboratory Assessments: Biochemistry: Alanine Aminotransferase (ALAT)
Description: Clinical laboratory assessments for ALAT at week 24 to end of trial visit.
Time Frame: Every 6th month, from week 24 to end of trial visit (week 173).
Population: The safety analysis set included all subjects who received at least one dose of the trial product.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | rFXIII 35 IU/kg
Number analyzed (Participants) | 6
IU/L
  Week 24 (pre-dose), N=4 | 17.75 (5.85)
  Week 48 (pre-dose), N=5 | 16.20 (2.39)
  Week 72 (pre-dose), N=5 | 16.40 (4.93)
  Week 96 (pre-dose), N=4 | 12.50 (3.70)
  Week 120 (pre-dose), N=3 | 21.33 (12.10)
  Week 144 (pre-dose), N=2 | 17.00 (1.41)
  Week 168 (pre-dose), N=1 | 14.00 (0.00)
  End of trial (week 173) pre-dose, N=5 | 16.00 (3.94)

6. Secondary Outcome: Clinical Laboratory Assessments: Biochemistry: Aspartate Aminotransferase (ASAT)
Description: Clinical laboratory assessments for ASAT at week 24 to end of trial visit.
Time Frame: Every 6th month, from week 24 to end of trial visit (week 173).
Population: The safety analysis set included all subjects who received at least one dose of the trial product.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | rFXIII 35 IU/kg
Number analyzed (Participants) | 6
IU/L
  Week 24 (pre-dose), N=4 | 30.75 (5.68)
  Week 48 (pre-dose), N=5 | 38.20 (10.99)
  Week 72 (pre-dose), N=5 | 31.20 (8.11)
  Week 96 (pre-dose), N=4 | 26.25 (1.71)
  Week 120 (pre-dose), N=3 | 27.00 (3.00)
  Week 144(pre-dose), N=2 | 26.00 (1.41)
  Week 168 (pre-dose), N=1 | 25.00 (0.00)
  End of trial (week 173) pre-dose, N=5 | 28.00 (3.61)

7. Secondary Outcome: Clinical Laboratory Assessments: Haematology: Haemoglobin
Description: Clinical values for haemoglobin collected from week 0 to end of trial visit.
Time Frame: Every 6th month, from week 0 to end of trial visit (week 173).
Population: The safety analysis set included all subjects who received at least one dose of the trial product.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | rFXIII 35 IU/kg
Number analyzed (Participants) | 6
mmol/L
  Week 0 (pre-dose), N=6 | 7.366 (0.25)
  Week 24 (pre-dose), N=4 | 7.624 (0.19)
  Week 48 (pre-dose), N=3 | 7.138 (0.31)
  Week 72 (pre-dose), N=3 | 7.262 (0.65)
  Week 96 (pre-dose), N=3 | 7.635 (0.27)
  Week 120 (pre-dose), N=3 | 7.821 (0.38)
  Week 144 (pre-dose), N=3 | 7.717 (0.70)
  Week 168 (pre-dose), N=2 | 7.759 (0.53)
  End of trial (week 173) pre-dose, N=6 | 8.048 (0.45)

8. Secondary Outcome: Clinical Laboratory Assessments: Haematology: Leucocytes
Description: Clinical laboratory values for leucocytes collected from week 0 to end of trial visit.
Time Frame: Every 6th month, from week 0 to end of trial visit (week 173).
Population: The safety analysis set included all subjects who received at least one dose of the trial product.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | rFXIII 35 IU/kg
Number analyzed (Participants) | 6
10^9 cells/L
  Week 0 (pre-dose), N=6 | 8.367 (2.20)
  Week 24 (pre-dose), N=4 | 7.373 (1.88)
  Week 48 (pre-dose), N=3 | 5.387 (1.06)
  Week 72 (pre-dose), N=4 | 5.863 (1.96)
  Week 96 (pre-dose), N=4 | 6.643 (1.89)
  Week 120(pre-dose), N=3 | 5.027 (2.12)
  Week 144(pre-dose), N=3 | 4.850 (3.00)
  Week 168(pre-dose), N=2 | 4.275 (2.65)
  End of trial (week 173) pre-dose, N=6 | 7.605 (1.25)

9. Secondary Outcome: Clinical Laboratory Assessments: Haematology: Thrombocytes
Description: Clinical laboratory values for thrombocytes collected from week 0 to end of trial visit.
Time Frame: Every 6th month, from week 0 to end of trial visit (week 173).
Population: The safety analysis set included all subjects who received at least one dose of the trial product.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | rFXIII 35 IU/kg
Number analyzed (Participants) | 6
10^9 cells/L
  Week 0 (pre-dose), N=6 | 316.3 (50.75)
  Week 24 (pre-dose), N=4 | 296.0 (54.17)
  Week 48 (pre-dose), N=3 | 277.0 (93.72)
  Week 72 (pre-dose), N=4 | 283.3 (41.63)
  Week 96 (pre-dose), N=4 | 332.3 (107.3)
  Week 120 (pre-dose), N=3 | 269.7 (102.2)
  Week 144 (pre-dose), N=3 | 324.3 (44.64)
  Week 168 (pre-dose), N=2 | 307.0 (15.56)
  End of trial (week 173) pre-dose, N=6 | 321.3 (60.45)

10. Secondary Outcome: Clinical Laboratory Assessments: Haematology: Erythrocytes
Description: Clinical laboratory values for erythrocytes collected from week 0 to end of trial visit.
Time Frame: Every 6th month, from week 0 to end of trial visit (week 173).
Population: The safety analysis set included all subjects who received at least one dose of the trial product.
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | rFXIII 35 IU/kg
Number analyzed (Participants) | 6
10^12 cells/L
  Week 0 (pre-dose), N=6 | 4.863 (0.43)
  Week 24 (pre-dose), N=4 | 4.745 (0.18)
  Week 48 (pre-dose), N=3 | 4.587 (0.12)
  Week 72 (pre-dose), N=4 | 4.505 (0.22)
  Week 96 (pre-dose), N=4 | 4.628 (0.26)
  Week 120 (pre-dose), N=3 | 4.247 (1.19)
  Week 144 (pre-dose), N=3 | 4.627 (0.11)
  Week 168 (pre-dose), N=2 | 4.875 (0.11)
  End of trial (week 173), N=6 | 4.662 (0.21)

11. Secondary Outcome: Clinical Laboratory Assessments: Haematology: Haematocrit
Description: Clinical laboratory values for haematocrit collected from week 0 to end of trial visit.
Time Frame: Every 6th month, from week 0 to end of trial visit (week 173).
Population: The safety analysis set included all subjects who received at least one dose of the trial product.
Measure: Mean (Standard Deviation); unit: percentage of red blood cells
Arm/Group | rFXIII 35 IU/kg
Number analyzed (Participants) | 6
percentage of red blood cells
  Week 0 (pre-dose), N=6 | 35.07 (0.99)
  Week 24 (pre-dose), N=4 | 36.05 (1.90)
  Week 48 (pre-dose), N=3 | 32.83 (1.76)
  Week 72 (pre-dose), N=4 | 34.80 (2.49)
  Week 96 (pre-dose), N=4 | 36.85 (1.07)
  Week 120 (pre-dose), N=3 | 32.83 (8.61)
  Week 144 (pre-dose), N=3 | 36.6 (3.44)
  Week 168 (pre-dose), N=2 | 36.40 (2.26)
  End of trial (week 173), N=6 | 37.45 (3.22)

12. Secondary Outcome: Physical Examinations
Description: Number of subjects in percentage with changes in values of physical examinations from week 0 to end of trial visit were collected.
Time Frame: Week 0 to end of trial visit (week 173).
Population: The safety analysis set included all subjects who received at least one dose of the trial product. Two abnormal physical examination findings related to skin and musculo-skeletal system were assessed as clinically significant by the investigator during the trial.
Measure: Number; unit: percentage of subjects
Arm/Group | rFXIII 35 IU/kg
Number analyzed (Participants) | 6
percentage of subjects
  Skin | 3
  Musculo-skeletal system | 1

13. Secondary Outcome: Vital Signs: Systolic BP (Blood Pressure)
Description: Values collected for systolic BP from week 0 to end of trial visit.
Time Frame: Week 0 to end of trial visit (week 173).
Population: The safety analysis set included all subjects who received at least one dose of the trial product.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | rFXIII 35 IU/kg
Number analyzed (Participants) | 6
mmHg
  Week 0, N=6 | 107.0 (13.7)
  Week 4, N=6 | 101.0 (8.4)
  Week 8, N=6 | 99.0 (9.4)
  Week 12, N=6 | 106.3 (9.4)
  Week 16, N=6 | 106.0 (4.1)
  Week 20, N=6 | 100.7 (10.0)
  Week 24, N=6 | 112.0 (12.6)
  Week 28, N=6 | 101.3 (11.4)
  Week 32, N=6 | 103.7 (20.6)
  Week 36, N=6 | 102.3 (11.9)
  Week 40, N=6 | 99.7 (8.3)
  Week 44, N=6 | 99.7 (13.0)
  Week 48, N=6 | 103.5 (19.4)
  Week 60, N=5 | 105.4 (7.8)
  Week 72, N=6 | 101.7 (7.3)
  Week 84, N=6 | 100.7 (10.7)
  Week 96, N=5 | 101.2 (4.8)
  Week 108, N=5 | 109.6 (10.9)
  Week 120, N=4 | 107.0 (7.0)
  Week 132, N=4 | 99.3 (6.2)
  Week 144, N=3 | 101.7 (7.8)
  Week 156, N=3 | 110.7 (7.0)
  Week 168, N=2 | 107.0 (7.1)
  End of trial (week 173), N=6 | 96.5 (4.8)

14. Secondary Outcome: Vital Signs: Diastolic BP (Blood Pressure)
Description: Values collected for diastolic BP from week 0 to end of trial visit.
Time Frame: Week 0 to end of trial visit (week 173).
Population: The safety analysis set one dose of the trial product.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | rFXIII 35 IU/kg
Number analyzed (Participants) | 6
mmHg
  Week 0, N=6 | 64.0 (7.6)
  Week 4, N=6 | 62.7 (11.4)
  Week 8, N=6 | 58.3 (19.1)
  Week 12, N=6 | 57.5 (7.9)
  Week 16, N=6 | 52.0 (3.3)
  Week 20, N=6 | 65.2 (6.5)
  Week 24, N=6 | 64.0 (4.4)
  Week 28, N=6 | 58.3 (10.4)
  Week 32, N=6 | 61.7 (16.4)
  Week 36, N=6 | 66.2 (11.1)
  Week 40, N=6 | 62.5 (6.4)
  Week 44, N=6 | 60.3 (7.3)
  Week 48, N=6 | 64.7 (10.9)
  Week 60, N=5 | 69.4 (10.9)
  Week 72, N=6 | 58.2 (4.6)
  Week 84, N=6 | 57.5 (8.1)
  Week 96, N=5 | 62.0 (6.3)
  Week 108, N=5 | 57.6 (10.4)
  Week 120, N=4 | 62.0 (3.4)
  Week 132, N=4 | 55.8 (8.4)
  Week 144, N=3 | 52.0 (9.2)
  Week 156, N=3 | 57.7 (6.7)
  Week 168, N=2 | 53.5 (2.1)
  End of trial (week 173), N=6 | 56.2 (5.5)

15. Secondary Outcome: Vital Signs: Pulse
Description: Values collected for pulse from week 0 to end of trial visit.
Time Frame: Week 0 to end of trial visit (week 173).
Population: The safety analysis included all subjects who received at least one dose of the trial product.
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | rFXIII 35 IU/kg
Number analyzed (Participants) | 6
beats/minute
  Week 0, N=6 | 113.2 (10.6)
  Week 4, N=6 | 97.7 (16.9)
  Week 8, N=6 | 106.2 (4.6)
  Week 12, N=6 | 104.5 (7.3)
  Week 16, N=6 | 109.8 (9.8)
  Week 20, N=6 | 105.3 (19.7)
  Week 24, N=6 | 103.7 (6.4)
  Week 28, N=6 | 102.2 (9.3)
  Week 32, N=6 | 108.3 (20.5)
  Week 36, N=6 | 95.5 (22.2)
  Week 40, N=6 | 93.2 (19.5)
  Week 44, N=6 | 95.5 (23.2)
  Week 48, N=6 | 100.5 (7.9)
  Week 60, N=5 | 109.0 (15.1)
  Week 72, N=6 | 100.8 (11.4)
  Week 84, N=6 | 99.3 (7.9)
  Week 96, N=4 | 96.5 (16.2)
  Week 108, N=5 | 98.4 (18.0)
  Week 120, N=4 | 85.0 (16.4)
  Week 132, N=4 | 86.3 (16.7)
  Week 144, N=3 | 88.0 (11.1)
  Week 156, N=3 | 100.7 (11.0)
  Week 168, N=2 | 92.0 (9.9)
  End of trial (week 173), N=6 | 94.0 (16.8)

16. Secondary Outcome: Rate (Number Per Subject Year) of All Bleeding Episodes Requiring Treatment With a FXIII Containing Product Other Than Recombinant Factor XIII.
Description: The rate (number per subject year) of all spontaneous, traumatic and intracranial bleeding episodes requiring treatment with FXIII-containing products during the rFXIII treatment period was assessed for treatment period.
Time Frame: Weeks 0 to end of trial visit (week 173).
Population: There were no bleeding episodes requiring treatment with a haemostatic agent (rFXIII) during the trial, which included subjects from full analysis set who received at least one dose of the trial product.
Arm/Group | rFXIII 35 IU/kg
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: All adverse events were collected and reported from screening (visit 1) and until the end of trial visit for a minimum period of 52 weeks.
Description: The safety analysis set included all subjects who received at least one dose of the trial product (rFXIII).
Arm/Group | rFXIII 35 IU/kg
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rFXIII 35 IU/kg (N=6)
Head injury (Injury, poisoning and procedural complications) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rFXIII 35 IU/kg (N=6)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (5)
Nausea (Gastrointestinal disorders) | 2 (2)
Tooth loss (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (4)
Fatigue (General disorders) | 1 (1)
Infusion site extravasation (General disorders) | 2 (2)
Infusion site rash (General disorders) | 1 (1)
Pain (General disorders) | 2 (2)
Pyrexia (General disorders) | 4 (6)
Acute tonsillitis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (3)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Otitis media acute (Infections and infestations) | 1 (2)
Pharyngitis streptococcal (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (7)
Varicella (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 3 (7)
Incorrect dose administered (Injury, poisoning and procedural complications) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (2)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 2 (2)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1)
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Bacterial test positive (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (7)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Snoring (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (3)
Haematoma (Vascular disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Limitations of the trial included the small number of subjects analysed and the sensitivity of the Berichrom® FXIII activity assay. However, congenital FXIII deficiency is a rare disease and there were no bleeds requiring haemostatic treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.